CLINICAL TRIAL: NCT00931853
Title: National Study, Phase III, Parallel, Double Blind, Placebo Comparative and Randomized to Evaluate the Therapeutic Efficacy and Tolerability of the Combination Naturetti® (Cassia Fistula + Senna Alexandrina Miller) in the Chronic Functional Constipation
Brief Title: Efficacy and Tolerability of Cassia Fistula Plus Senna Alexandrina Miller (Sugar Free) in the Chronic Functional Constipation (CFC).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENCA_L_04392
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

ARMS (1):
- SENNA + CASSIA (Naturetti) (Experimental): Daily administration (oral) of one spoon (5g) of Naturetti (SENNA+CASSIA) jelly sugar free at bedtime, during 30 days
  Interventions: Drug: SENNA+CASSIA(Naturetti)

INTERVENTIONS:
Drug: SENNA+CASSIA(Naturetti) — Daily administration (oral) of one spoon (5g) of Naturetti (SENNA+CASSIA) jelly sugar free at bedtime, during 30 days

SUMMARY:
Primary Objective:

* To evaluate the clinical efficacy of Naturetti (jelly sugar free)
* To test medication on subjects who suffer chronic functional constipation in 30 days use.

Secondary Objectives:

* To demonstrate the clinical tolerability when daily used (repeated doses) of the components of the study drug. The components will be evaluated by the adverse events occurrence classified by possibly related, probably related and definitely related
* To demonstrate the clinical tolerability of the study medication by the continuous use during the second phase study
* To identify any adverse events related to the study drug
* To identify any drug interaction.

ELIGIBILITY:
Inclusion criteria:

* Having chronic functional constipation by ROME IIII criteria
* Having the majority of the stool as type 1 or 2 by Bristol Stool Scale
* Female subjects should be using an effective contraceptive method more than 3 months if they are sexually active and on reproductive stage
* ICF signature
* Be able to understand and agree to undertake the study procedures
* Having no contraindication related to the study drug
* To perform all study visits.

Exclusion criteria:

* Having previous history or current neurological disorder and/or metabolic one
* Having constipation caused by previous surgery
* Having intestinal obstruction including colon/rectum cancer
* Having endocrine disorder as diabetes mellitus
* Having Irritable bowel syndrome or inflammatory bowel disease
* Having multiple sclerosis
* Having Parkinsons disease
* Having Hirschsprungs disease and dyssynergy defecation
* Continuous treatment with the following: analgesics, anticholinergic (antihistamines, antispasmodics, antidepressants, antipsychotics) iron supplements or aluminum, opiates, antihypertensive, calcium channel blockers and ganglionic blocker
* Treatment with any other laxative medication other than the rescue medication during the study
* Patients who could not confirm the chronic functional constipation during the phase I study
* Pregnancy or breast feeding woman
* Abnormal laboratory results, or clinical result that shows significant by the Investigator
* Corporeal mass index > 30
* Patients who have participate in other clinical study within 30 days
* Unable to fulfill the questionnaire (diary)
* Any condition that makes impossible to the patient in participates by Investigator opinion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Measure of the chronic functional constipation symptoms based on the Rome III criteria | From the baseline to the end of the study (at 30 days)

SECONDARY OUTCOMES:
Evaluation of the stool aspect based on the Bristol Stool Scale | From the baseline to the end of the study (at 30 days)
Evaluation of the use of sene extract as rescue medication | From the baseline to the end of the study (at 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil